CLINICAL TRIAL: NCT00616486
Title: A Multicentre, Double-blind, Randomized, Placebo-controlled Study Evaluating the Efficacy, Safety, and Clinical Outcomes of Low Frequency, Repetitive Transcranial Magnetic Stimulation (Over Supplementary Motor Area (SMA) Applied Bilaterally and Simultaneously) Versus Sham (Placebo rTMS) Treatment for 6 Weeks, When Added to a Stable Pharmacotherapy in Subjects With Obsessive Compulsive Disorder (OCD).
Brief Title: rTMS in Treatment of Obsessive Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Military Medical Academy, Bulgaria (Other); Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Dr. Roumen Milev, Professor of Psychiatry and Psychology, Head, Department of Psychiatry Queen's University, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: psiy-266-07
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation
- 2 (Placebo Comparator)
  Interventions: Device: sham (placebo)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — 6 weeks of stimulation with RMT frequency 1Hz, intensity 110% of RMT for 20 minutes, 5 minutes of trains with 2 minutes of intra-train intervals to both SMA. Treatment will be given 5 times a week for 4 weeks, 3 times a week during Week 5 and 2 times a week during Week 6.
  Other Names: rTMS machine (MagPro, Medtronic)
  Arms: 1
Device: sham (placebo) — Sham treatment will mimic active treatment mentioned above.
  Other Names: rTMS machine (MagPro, Medtronic).
  Arms: 2

SUMMARY:
Low frequency (1Hz) rTMS applied bilaterally and simultaneously over SMA for 6 weeks in addition to the standard treatment regimen for OCD, will lead to significant improvement in patients' symptoms. The clinical improvement detected by YBOCS, CGI and SF-36 QOLS scores will be statistically significant in active treatment group compared to sham (placebo) treatment group.

ELIGIBILITY:
Inclusion Criteria:

* signed patient informed consent;
* primary obsessive compulsive disorder;
* YBOCS score at least 20;
* males/females 18-65yrs;
* treated with adequate dose of SSRI at least 8 weeks at some stage of illness;
* currently using adequate, stable dose of SSRI at least 4 weeks but not responding.

Exclusion Criteria:

* schizophrenia, other psychotic disorders, bipolar I, current major depressive disorder (HDRS(17)>18, substance/alcohol dependence within last 6 months;
* severe axis II;
* suicidal score>=6 on MINI;
* metallic implant in cranium;
* severe/unstable medical conditions;
* not responding to ECT or had TMS in last 6 months;
* history epilepsy;
* neurological disorder leading to increased intracranial pressure;
* severe cardiac disorder/intracardiac lines, pacemakers;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (YBOCS) | pre, week 1, 2, 4, 6, 8, 12

SECONDARY OUTCOMES:
Clinical Global Impression | pre, week 1, 2, 4, 6, 8, 12
Hamilton Depression Rating Scale-21(HDRS) | pre, week 1, 2, 4, 6, 8, 12
Pittsburgh Sleep Quality Index (PSQI) | pre, week 1, 2, 4, 6, 8, 12
Hamilton Anxiety Rating Scale (HARS) | pre, week 1, 2, 4, 6, 8, 12
SF-36 QOLS version (1) | pre, week 1, 2, 4, 6, 8, 12
Visual Analogue Scale | pre, week 1, 2, 4, 6, 8, 12

CONTACTS AND LOCATIONS:
Overall Officials: Roumen Milev, MD, Study Chair — Queen's University
Locations (3):
- Military Medical Academy, Sofia, Bulgaria
- Providence Care, Mental Health Services, Kingston, Ontario, Canada
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Hawken ER, Dilkov D, Kaludiev E, Simek S, Zhang F, Milev R. Transcranial Magnetic Stimulation of the Supplementary Motor Area in the Treatment of Obsessive-Compulsive Disorder: A Multi-Site Study. Int J Mol Sci. 2016 Mar 22;17(3):420. doi: 10.3390/ijms17030420. PMID 27011177